CLINICAL TRIAL: NCT02340234
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Lebrikizumab in Patients With Persistent Moderate to Severe Atopic Dermatitis That is Inadequately Controlled by Topical Corticosteroids
Brief Title: A Study of Lebrikizumab in Participants With Persistent Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS29250; 2014-000049-56 (EudraCT Number)
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Lebrikizumab 250 mg Single Dose + TCS Cream (Experimental): Participants will receive lebrikizumab 250 milligrams (mg) SC single dose on Day 1 followed by placebo on Week 4 and Week 8. Participants will continue to apply TCS cream (triamcenolone acetonide 0.1% or hydrocortisone 2.5% cream) twice daily to active skin lesions throughout the 12-week treatment period.
  Interventions: Drug: Lebrikizumab; Drug: Placebo; Drug: TCS Cream
- Lebrikizumab 125 mg Single Dose + TCS Cream (Experimental): Participants will receive lebrikizumab 125 mg SC single dose on Day 1 followed by placebo on Week 4 and Week 8. Participants will continue to apply TCS cream (triamcenolone acetonide 0.1% or hydrocortisone 2.5% cream) twice daily to active skin lesions throughout the 12-week treatment period.
  Interventions: Drug: Lebrikizumab; Drug: Placebo; Drug: TCS Cream
- Lebrikizumab 125 mg Q4W + TCS Cream (Experimental): Participants will receive lebrikizumab 125 mg SC every 4 weeks (Q4W) for a total of 3 doses. Participants will continue to apply TCS cream (triamcenolone acetonide 0.1% or hydrocortisone 2.5% cream) twice daily to active skin lesions throughout the 12-week treatment period.
  Interventions: Drug: Lebrikizumab; Drug: TCS Cream
- Placebo Q4W + TCS Cream (Placebo Comparator): Participants will receive placebo Q4W for a total of 3 doses. Participants will continue to apply TCS cream (triamcenolone acetonide 0.1% or hydrocortisone 2.5% cream) twice daily to active skin lesions throughout the 12-week treatment period.
  Interventions: Drug: Placebo; Drug: TCS Cream

INTERVENTIONS:
Drug: Lebrikizumab — Lebrikizumab will be administered SC as per the schedule specified in the respective arms.
  Arms: Lebrikizumab 125 mg Q4W + TCS Cream; Lebrikizumab 125 mg Single Dose + TCS Cream; Lebrikizumab 250 mg Single Dose + TCS Cream
Drug: Placebo — Placebo matching to lebrikizumab will be administered as per the schedule specified in the respective arms.
  Arms: Lebrikizumab 125 mg Single Dose + TCS Cream; Lebrikizumab 250 mg Single Dose + TCS Cream; Placebo Q4W + TCS Cream
Drug: TCS Cream — TCS cream (triamcenolone acetonide 0.1% or hydrocortisone 2.5% cream) twice daily

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the safety and efficacy of lebrikizumab administered subcutaneously (SC) in adult participants with persistent moderate to severe atopic dermatitis (AD) who are inadequately controlled by topical corticosteroids (TCS). The study includes a screening visit, a 2-week run-in period, a 12-week blinded treatment period, and an 8-week safety follow-up period. Following screening visit, eligible participants will enter in run-in period (Days - 14 to - 1) during which a protocol-specified topical therapy regimen will be initiated. At the end of the run-in period, participants who have: 1) demonstrated compliance with the protocol-specified TCS regimen, and 2) who continue to fulfill the eligibility criteria will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* AD diagnosed by the Hanifin/Rajka criteria and that has been present for at least 1 year at screening
* Moderate to severe AD as graded by the Rajka/Langeland criteria at screening
* History of inadequate response to a >/= 1 month (within the 3 months prior to the screening visit) treatment regimen of at least daily TCS and regular emollient for treatment of AD
* EASI score >/= 14 at screening and end of the run-in period
* IGA score >/= 3 (5-point scale) at screening and end of the run-in period
* AD involvement of >/= 10% BSA at screening
* Pruritus VAS score >/= 3 at screening

Exclusion Criteria:

* Past and/or current use of any anti-interleukin (IL)-13 or anti-IL-4/IL-13 therapy, including lebrikizumab
* Use of an investigational agent within 4 weeks prior to screening or within 5 half-lives of the investigational agent, whichever is longer
* History of a severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the lebrikizumab injection
* Use of any complementary, alternative, or homeopathic medicines including, but not limited to, phytotherapies, traditional or non-traditional herbal medications, essential fatty acids, or acupuncture within 7 days prior to the run-in period or need for such medications during the study
* Evidence of other skin conditions; including, but not limited to, T-cell lymphoma or allergic contact dermatitis
* Evidence of, or ongoing treatment (including topical antibiotics) for active skin infection at screening
* Other recent infections meeting protocol criteria
* Active tuberculosis requiring treatment within the 12 months prior to Visit 1
* Evidence of acute or chronic hepatitis or known liver cirrhosis
* Known immunodeficiency, including human immunodeficiency virus (HIV) infection
* Use of a topical calcineurin inhibitor (TCI) at the time of screening, unless the participant is willing to stop TCI use during the study (including the run-in period) and, in the investigator's opinion, it is safe to do so
* Clinically significant abnormality on screening electrocardiogram (ECG) or laboratory tests that, in the opinion of the investigator, may pose an additional risk in administering study drug or TCS to the participant
* Known current malignancy or current evaluation for a potential malignancy, including basal or squamous cell carcinoma of the skin or carcinoma in situ
* History of malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a 50 Percent (%) Reduction From Baseline in Eczema Area and Severity Index (EASI) Score (EASI-50) at Week 12 | Week 12

SECONDARY OUTCOMES:
Percent Change From Baseline in EASI Score at Week 12 | Baseline, Week 12
Absolute Change From Baseline in EASI Score at Week 12 | Baseline, Week 12
Percentage of Participants Achieving a 75% Reduction From Baseline in EASI Score (EASI-75) at Week 12 | Week 12
Percentage of Participants Achieving an Investigator's Global Assessment (IGA) score of 0 or 1 at Week 12 | Week 12
Percentage of Participants With a Greater Than or Equal to (>/=) 2 Point Reduction From Baseline in IGA at Week 12 | Week 12
Absolute Change From Baseline in IGA at Week 12 | Baseline, Week 12
Percentage of Participants Achieving an Investigator Global Signs Assessment (IGSA) Score of 0 or 1 at Week 12 | Week 12
Percentage of Participants with a >/=2 Point Reduction From Baseline in IGSA at Week 12 | Week 12
Absolute Change From Baseline in IGSA at Week 12 | Baseline, Week 12
Percent Change From baseline in Severity Scoring of Atopic Dermatitis (SCORAD) at Week 12 | Baseline, Week 12
Absolute Change From baseline in SCORAD at Week 12 | Baseline, Week 12
Percentage of Participants With a 50% or 75% Reduction From Baseline in SCORAD-50/75 at Week 12 | Week 12
Percentage of Participants Achieving EASI-50 at Week 12 and Maintaining EASI-50 at Weeks 16 | Weeks 12, 16
Percentage of Participants Achieving EASI-50 at Week 12 and Maintaining EASI-50 at Weeks 16 and 20 | Weeks 12, 16, 20
Percentage of Participants Achieving IGA Score of 0 or 1 at Week 12 and Maintaining IGA Score of 0 or 1 at Weeks 16 | Weeks 12, 16
Percentage of Participants Achieving IGA Score of 0 or 1 at Week 12 and Maintaining IGA Score of 0 or 1 at Weeks 16 and 20 | Weeks 12, 16, 20
Percentage of Participants Achieving IGSA Score of 0 or 1 at Week 12 and Maintaining IGSA Score of 0 or 1 at Weeks 16 | Weeks 12, 16
Percentage of Participants Achieving IGSA Score of 0 or 1 at Week 12 and Maintaining IGSA Score of 0 or 1 at Weeks 16 and 20 | Weeks 12, 16, 20
Percentage of Participants Achieving SCORAD-50 at Week 12 and Maintaining SCORAD-50 at Weeks 16 | Weeks 12, 16
Percentage of Participants Achieving SCORAD-50 at Week 12 and Maintaining SCORAD-50 at Weeks 16 and 20 | Weeks 12, 16, 20
Percent Change From Baseline in Total % Body Surface Area (BSA) Affected At Week 12 | Baseline, Week 12
Absolute Change From Baseline in Pruritus as Measured by the Pruritus Visual Analog Scale (VAS) at Week 12 | Baseline, Week 12
Percent Change From Baseline in Pruritus as Measured by the Pruritus VAS at Week 12 | Baseline, Week 12
Absolute Change From Baseline in Pruritus as Measured by the 5-D Itch Scale at Week 12 | Baseline, Week 12
Percent Change From Baseline in Pruritus as Measured by the 5-D Itch Scale at Week 12 | Baseline, Week 12
Total Use (Grams) of TCS From Baseline to Week 12 | From Baseline to Week 12
Total Use (Grams) of TCS From Week 12 to End of Study or Early Termination | From Week 12 to end of study or early termination (up to approximately 20 weeks)
Number of Disease Flares From Baseline to Week 12 | From Baseline to Week 12
Change in AD Symptoms From Baseline to Week 12, as Assessed by the Atopic Dermatitis Symptom Diary (ADSD) | Baseline, Week 12
Change in AD-Specific HealthRelated Quality of Life (QoL) From Baseline to Week 12, as Assessed by the Atopic Dermatitis Impact Questionnaire (ADIQ) | Baseline, Week 12
Change in Health-Related QoL From Baseline to Week 12, as Measured by the Dermatology Life Quality Index (DLQI) | Baseline, Week 12
Percentage of Participants With Treatment-Emergent Adverse Events (AEs) | From start of run-in period (Day -14) until study completion (up to approximately 20 Weeks)
Percentage of Participants With Anti-Therapeutic Antibodies (ATA) to Lebrikizumab | Pre-dose on Days 1, 29, 85, 141, study discontinuation visit (up to Day 141)
Percentage of Participants With ATA to Phospholipase B-Like 2 (PLBL2) Protein | Pre-dose on Days 1, 29, 85, 141, study discontinuation visit (up to Day 141)
Percentage of Participants With Disease Rebound | From Week 12 up to approximately 20 weeks
Maximum Serum Concentration (Cmax) of Lebrikizumab | After first dose of lebrikizumab at Week 1
Time to Reach Cmax (Tmax) of Lebrikizumab | After first dose of lebrikizumab at Week 1
Minimum Serum Concentration (Cmin) of Lebrikizumab | Pre-dose at Weeks 4, 8, 12
Elimination Half-Life (t1/2) of Lebrikizumab | Pre-dose on Days 1, 8, 29, 43, 57, 85, 113, 141, study discontinuation visit (up to Day 141)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (74):
- United States (16):
  - Dermatology Research Associate, Los Angeles, California
  - UCSD Division of Dermatology, San Diego, California
  - Univ of Calif-San Francisco, San Francisco, California
  - University of Colorado; Anschutz Cancer Pavilion, Aurora, Colorado
  - Ameriderm Research, Ormond Beach, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - University of Iowa Healthcare; Dermatology, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Somerset Skin Centre, Troy, Michigan
  - Washington University; Dermatology, St Louis, Missouri
  - Sadick Research Group, New York, New York
  - Oregon Health & Science University; Department of Dermatology, Portland, Oregon
  - University of Texas Medical School-Houston, Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Virginia Clinical Research Inc., Norfolk, Virginia
- Australia (4):
  - St George Dermatology and Skin Cancer Centre, Kogarah, New South Wales
  - Skin & Cancer Foundation, Carlton, Victoria
  - Royal Melbourne Hospital; Dermatology Department, Parkville, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
- Canada (7):
  - Institute for Skin Advancement, Calgary, Alberta
  - Guildford Dermatology Specialists, Surrey, British Columbia
  - Dr. Melinda Gooderham Medicine Professional Corporation, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
  - XLR8 Medical Research Inc., Windsor, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
- Czechia (3):
  - Faculty Hospital; Department of Dermatology, Pilsen
  - Charles University School of Medicine; Deptartment of Dermatology, Prague
  - Masarykova nemocnice o.z; kozni oddeleni, Ústí nad Labem
- Finland (3):
  - Helsinki University Central Hospital; Skin & Allergy Hospital, Helsinki
  - Tampere University Hospital; Dermatology and allergology, Tampere
  - Turku Central University Hospital; Dermatology and allergology, Turku
- France (5):
  - Hopital Saint Andre CHU De Bordeaux; Dermatologie, Bordeaux
  - Hopital du Bocage; Dermatologie, Dijon
  - Hopital Hotel Dieu Et Hme; Clinique Dermatologique, Nantes
  - Hopital l Archet 2; Ginestriere, Service de; Dermatologie, Nice
  - Centre Hospitalier Lyon Sud; Dermatologie, Pierre-Bénite
- Germany (6):
  - Charite Mitte; Klinik fur Dermatologie, Berlin
  - Universitätsklinik Bonn, Bonn
  - Klinik Johann Wolfgang von Goethe Uni; Klinik für Dermatologie, Venerologie und Allergologie, Frankfurt
  - SRH Wald-Klinikum Gera GmbH; Hautkrankheiten und Allergologie, Gera
  - UKSH Kiel; Klinik für Dermatologie, Venerologie und Allergologie, Kiel
  - Universitätsklinikum Mainz, Mainz
- Netherlands (3):
  - Academisch Medisch Centrum Universiteit Amsterdam; Dermatology and VU University Medical Center, Amsterdam
  - University Medical Center Groningen; Department of Dermatology, Groningen
  - UMC Utrecht; Dermatology, Utrecht
- Poland (5):
  - Uniwersyteckie Centeum Kliniczne GUMed; Klinika Dermatologii, Wenerologii i Alergologii, Gdansk
  - DERMED Centrum Medyczne; Sp zoo, Lodz
  - Laser Clinic, Szczecin
  - ALERGO-MED Specjalistyczna Przychodnia Lekarska Sp. z o. o, Tarnów
  - dermMedica sp.z o.o., Wroclaw
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - ChungAng University Hospital, Seoul
- Spain (7):
  - Clinica Universitaria de Navarra; Servicio de Dermatologia, Pamplona, Navarre
  - Hospital de la Santa Creu i Sant Pau; Servicio de Dermatologia, Barcelona
  - Hospital Universitario La Princesa, Servicio dermatologia, Madrid
  - HUGregorio Marañón, Servicio de dermatología, Madrid
  - Hospital Ramon y Cajal; servicio dermatologia, Madrid
  - Hospital Universitario La Paz; Servicio de dermatologia, Madrid
  - Hospital General Universitario de Valencia; servicio de dermatología, Valencia
- Switzerland (3):
  - Inselspital Bern; Dermatologie, Bern
  - CHUV; Dermatologie, Lausanne
  - Universitätsspital Zürich; Dermatologische Klinik, Zurich
- Taiwan (3):
  - Chang Gung Medical Foundation;Kaohsiung Branch; Department of Dermatology, Kaohsiung City
  - National Cheng-Kung University Hospital; Department of Dermatology, Tainan
  - National Taiwan University Hospital; Department of Dermatology, Taipei
- United Kingdom (6):
  - Russells Hall Hospital, Dudley
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital; Skin Therapy Research Unit, London
  - Newcastle University & The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Churchill Hospital, Oxford
  - Poole Hospital, Poole
  - Salford Royal NHS Foundation Trust, Salford